CLINICAL TRIAL: NCT03251222
Title: Intranasal Sedation With Dexmedetomidine for Vitroretinal Procedures
Brief Title: Intranasal Sedation With Dexmedetomidine
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Iztok Potocnik, M.D., PHD, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UKC-OCKL1
Record Dates: First submitted 2017-08-02; First posted 2017-08-16 (Actual); Last update posted 2017-08-16 (Actual); Status verified 2017-08

CONDITIONS: Conscious Sedation
Keywords: conscious sedation, vitroretinal procedures
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexmedetomidine group (Experimental): Patients who will receive Dexmedetomidine intranasal prior the sedation with remifentanil
  Interventions: Drug: Dexmedetomidine
- Placebo Concentrate (Placebo Comparator): Patients will recive 0.9% NaCl
  Interventions: Other: Placebo - Concentrate

INTERVENTIONS:
Drug: Dexmedetomidine — Intranasal aplication of dexmedetomidine
  Arms: Dexmedetomidine group
Other: Placebo - Concentrate — Intranasal aplication of 0.9% NaCl
  Other Names: Placebo
  Arms: Placebo Concentrate

SUMMARY:
For patients with eye surgery and shorter surgery, sedation is a well-established method in preserved consciousness and has been successfully used for several years. We have also developed and published a valid protocol (1).

Remifentanil is used in intravenous infusion for sedation and anxiolysis. Remifentanil is a descriptive analgesic, which also works partially anxiolytically. In eye surgery, it is important that the patient cooperates during the operation and should not be ashamed, as injury to the eye could occur, because the vitrectomes are performed with a fine intraocular endoscopic technique, in which the operator inserts his instruments through the whiteness into the eye. For this reason, we have not yet added additional sedatives (for example, midazolam), which is very unpredictable as regards sedation. Remifentanil is also very unpredictable and it is very difficult to control it during the operation so that the patient is saturated with satisfaction.

Lately, dexmedetomidine has been successfully used in sedation for other areas of surgery (eg neurosurgery, maxillofacial surgery, ORL). It is a safe, proven, active substance with alpha 2 agonistic effect, which has not yet been used in the field of ocular surgery and has not yet published articles in this field. The substance is very suitable because it works mildly sedative and at the same time analgesic.

DETAILED DESCRIPTION:
For patients with eye surgery and shorter surgery, sedation is a well-established method in preserved consciousness and has been successfully used for several years. We have also developed and published a valid protocol (1).

Remifentanil is currently used for intravenous infusion for analgesia and anxiolysis. Remifentanil is an opioid analgesic, which also works partially anxiolytically. It has been studied in detail for postnatal analgesia (2). In eye surgery, it is important that the patient cooperates during the operation and should not be ashamed, as injury to the eye could occur, because the vitrectomes are performed with a fine intraocular endoscopic technique, in which the operator inserts his instruments through the whiteness into the eye. For this reason, we have not yet added additional sedatives (for example, midazolam), which is very unpredictable and a rapidly shallow sedation can pass into the deeper. Remifentanil is also very unpredictable and it is very difficult to control it during the operation, so that the patient is satisfactorily analgesized at all times, but still co-operable.

Recently, dexmedetomidine (3-5) has been successfully used in other areas of surgery (eg neurosurgery, maxillofacial surgery, ORL) and intensive sedation therapies. It is a safe, proven, active substance with alpha 2 agonistic effect, which has not yet been used in the field of ocular surgery and has not yet published articles in this field. The substance is very suitable because it works mildly sedative and at the same time analgesic (3).

Dexmedetomidine is predominantly administered intravenously, and intranasal administration (6-8) has also been established in pediatric patients.

We decided to use intranasal use because it is simple, safe and suitable for such treatments because intravenous dexmedetomidine could not be administered because it should be given enough time before surgery (at least 40 min) because otherwise the appropriate effect . Patients for such operations will enter the operating room directly from the departments on foot and dexmedetomidine could not be started earlier, as it is not possible to provide adequate control in the department. A sedentary patient would also not be able to walk into an operational one, which would greatly complicate and also increase logistics.

The study is applicable, as it will provide objective indicators, which type of sedation is most effective and safe for vitreoretinal interventions.

ELIGIBILITY:
Inclusion Criteria: patients who will be operated on the eye (vitreoretinal interventions) patients with ASA status 1-3

-

Exclusion Criteria:

* patients who will not want to be operated in the sedation but in general anesthesia
* poor general condition (ASA> 3)
* with severe cardiac disease (NYHA> 3)
* with severe pulmonary obstructive disease (FEV1 <40%)
* neurological diseases
* psychiatric patients
* patients receiving regular psychotropic treatment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-12-01 (Estimated); Study Completion 2018-03-01 (Estimated)

PRIMARY OUTCOMES:
remifentanil consuption | duration of the procedure
  the consuption of remifentanil requiered to reach the appropriate sedation will be meassured

SECONDARY OUTCOMES:
Oxigen Saturation | duration of the procedure
  Oxigen Saturation measured with pulse oxymetry

OTHER OUTCOMES:
BIS- bispectral index | duration of the procedure
  Depth of the sedation

CONTACTS AND LOCATIONS:
Overall Officials: Vesna Novak-Jankovic, PROF, Study Chair — UMCLjubljana, KOAIT
Locations (1):
- UMCLjubljana, CD of Anaesthesiology and Intensive Therapy, Ljubljana, Slovenia

REFERENCES:
- [Result] Ohashi Y, Baghirzada L, Sumikura H, Balki M. Erratum to: Remifentanil for labor analgesia: a comprehensive review. J Anesth. 2017 Feb;31(1):160. doi: 10.1007/s00540-016-2269-z. No abstract available. PMID 27770212
- [Result] Das S, Al-Mashani A, Suri N, Salhotra N, Chatterjee N. Combination of Continuous Dexmedetomidine Infusion with Titrated Ultra-Low-Dose Propofol-Fentanyl for an Awake Craniotomy. Sultan Qaboos Univ Med J. 2016 Aug;16(3):e347-51. doi: 10.18295/squmj.2016.16.03.014. Epub 2016 Aug 19. PMID 27606116
- [Result] Martinez-Simon A, Cacho-Asenjo E, Hernando B, Honorato-Cia C, Naval L, Panadero A, Nunez-Cordoba JM. Loading dose of Dexdor(R) and optimal sedation during oral and maxillofacial ambulatory surgery procedures: An observational study. Rev Esp Anestesiol Reanim. 2017 Apr;64(4):206-213. doi: 10.1016/j.redar.2016.08.005. Epub 2016 Nov 5. English, Spanish. PMID 27825666
- [Result] Xu J, Deng XM, Yang D, Wei LX, Zhi J, Xu WL, Liu JH. Comparison of Sedative Effects of Two Spray Administration of Intranasal Dexmedetomidine Doses for Premedication in Children. Zhongguo Yi Xue Ke Xue Yuan Xue Bao. 2016 Oct 10;38(5):563-567. doi: 10.3881/j.issn.1000-503X.2016.05.013. PMID 27825415
- [Result] Ghai B, Jain K, Saxena AK, Bhatia N, Sodhi KS. Comparison of oral midazolam with intranasal dexmedetomidine premedication for children undergoing CT imaging: a randomized, double-blind, and controlled study. Paediatr Anaesth. 2017 Jan;27(1):37-44. doi: 10.1111/pan.13010. Epub 2016 Oct 13. PMID 27734549
- [Result] Bonanno LS, Pierce S, Badeaux J, FitzSimons JJ. Effectiveness of preoperative intranasal dexmedetomidine compared with oral midazolam for the prevention of emergence delirium in pediatric patients undergoing general anesthesia: a systematic review protocol. JBI Database System Rev Implement Rep. 2016 Aug;14(8):70-9. doi: 10.11124/JBISRIR-2016-003059. PMID 27635747